CLINICAL TRIAL: NCT01991873
Title: Randomized Phase II Study for Evaluation of Efficacy and Safety of Maintenance Treatment With 5-FU/FA Plus Panitumumab vs. 5-FU/FA Alone After Prior Induction Treatment With mFOLFOX6 Plus Panitumumab and Re-induction With mFOLFOX6 Plus Panitumumab in Case of Progression for First-line Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Maintenance Therapy With 5-FU/FA Plus Panitumumab vs. 5-FU/FA Alone After Prior Induction and Re-induction After Progress for 1st-line Treatment of Metastatic Colorectal Cancer
Acronym: PanaMa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: ClinAssess GmbH (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0212; 2012-005422-30 (EudraCT Number); PanaMa_DE-2009-0003 (Other: Amgen)
Record Dates: First submitted 2013-10-22; First posted 2013-11-25 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; maintenance therapy; Panitumumab; Vectibix®
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Maintenance Chemotherapy; Leucovorin; Fluorouracil; Panitumumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance Chemotherapy + Panitumumab (Experimental): Maintenance therapy:
  Panitumumab 6 mg/kg prior to administration of chemotherapy Folinic acid 400 mg/m2 over 2 hours on day 1 5-FU 2400mg/m2 46h continuous infusion day 1 - day 2 Repeat on day 15
  Re-induction upon progression:
  Panitumumab 6 mg/kg prior to administration of mFOLFOX6 chemotherapy.
  mFOLFOX6: Oxaliplatin 85 mg/m2 over 2 hours on day 1 Folinic acid 400 mg/m2 over 2 hours on day 1 5-FU 2400mg/m2 46h continuous infusion day 1 - day 2 Repeat on day 15
  Interventions: Drug: Maintenance Chemotherapy; Drug: Panitumumab (Within maintenance phase); Drug: mFOLFOX6 (Within re-induction phase); Drug: Panitumumab (Within re-induction phase)
- Maintenance Chemotherapy w/o Panitumumab (Experimental): Maintenance therapy:
  Folinic acid 400 mg/m2 over 2 hours on day 1 5-FU 2400mg/m2 46h continuous infusion day 1 - day 2 Repeat on day 15
  Re-induction upon progression:
  Panitumumab 6 mg/kg prior to administration of mFOLFOX6 chemotherapy.
  mFOLFOX6 chemotherapy: Oxaliplatin 85 mg/m2 over 2 hours on day 1 Folinic acid 400 mg/m2 over 2 hours on day 1 5-FU 2400mg/m2 46h continuous infusion day 1 - day 2 Repeat on day 15
  Interventions: Drug: Maintenance Chemotherapy; Drug: mFOLFOX6 (Within re-induction phase); Drug: Panitumumab (Within re-induction phase)

INTERVENTIONS:
Drug: Maintenance Chemotherapy
  Other Names: Folinic acid + 5-FU (5-Fluorouracil)
Drug: Panitumumab (Within maintenance phase)
  Other Names: Vectibix
  Arms: Maintenance Chemotherapy + Panitumumab
Drug: mFOLFOX6 (Within re-induction phase)
  Other Names: Oxaliplatin + Folinic acid + 5-FU (5-Fluorouracil)
Drug: Panitumumab (Within re-induction phase)
  Other Names: Vectibix

SUMMARY:
This is a phase II, randomized, multi-center, open-label, parallel-group study to evaluate the progression-free survival during maintenance therapy.

Eligible patients will be treated within a 12-week induction therapy. Those patients achieving CR/PR or SD at 12 weeks and qualifying for maintenance treatment and re-induction treatment with all potential drug components, will be randomized in a ratio of 1:1 to receive chemotherapy plus panitumumab or chemotherapy alone during maintenance. In case of progression, re-induction treatment will be started.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female ≥ 18 years of age
* Histologically proven metastatic colorectal cancer
* Molecular testing showing RAS wild-type in colorectal carcinoma cells
* Life expectancy > 12 weeks
* At least one measurable lesion according to RECIST 1.1
* Adequate bone marrow, liver, kidney, organ and metabolic function
* Bone marrow function:

  * leukocyte count ≥ 3.0 × 109/L
  * ANC ≥ 1.5 × 109/L
  * platelet count ≥ 100 × 109/L
  * hemoglobin ≥ 9 g/dL or 5.59 mmol/L (may be transfused or treated with erythropoietin to maintain/ exceed this level)
* Hepatic function:

  * Total bilirubin ≤ 1.5 × UNL
  * ALT and AST ≤ 2.5 × UNL (or ≤ 5 × UNL in presence of liver metastases)
  * AP ≤ 5 × UNL
* Renal function:

  * Creatinine clearance ≥ 50 mL/min according to Cockcroft-Gault formula or serum creatinine ≤ 1.5 × UNL
* Metabolic function:

  * Magnesium ≥ lower limit of normal
  * Calcium ≥ lower limit of normal
* ECOG performance status 0 - 1
* Women of child-bearing potential must have a negative pregnancy test

Exclusion Criteria:

* Previous treatment for colorectal cancer in the metastatic setting
* Previous EGFR-targeting therapy < 6 months after end of adjuvant therapy
* Known brain metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and steroids
* Chronic inflammatory bowel disease
* Peripheral neuropathy ≥ NCI-CTCAE V 4.03 grade 2
* Other previous malignancies with the exception of a history of previous curatively treated basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix or other curatively treated malignant disease without recurrence after at least 5 years of follow-up
* Significant disease that, in the investigator's opinion, would exclude the patient from the study
* History of cardiac disease; defined as:

  * Congestive heart failure > New York Heart Association (NYHA) class 2
  * Active coronary artery disease (myocardial infarction more than 6 months prior to start of study treatment is allowed)
  * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted)
  * Uncontrolled hypertension (defined as blood pressure ≥ 160 mmHg systolic and/or ≥ 90 mmHg diastolic on medication)
* Patients with interstitial lung disease, e.g., pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Known HIV, hepatitis B or C infection
* Known hypersensitivity reaction to any of the study components
* Radiotherapy, major surgery or any investigational drug 30 days before registration
* Pregnancy or lactation or planning to be pregnant during treatment and within 6 months after the end of treatment
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for at least an additional 6 months after the end of treatment
* Known alcohol or drug abuse
* Any condition that is unstable or could jeopardize the safety of the patient and his compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2014-04; Primary Completion 2023-02-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Until end of follow-up (24 months after randomization)
  Progression-free survival during maintenance therapy defined as time from randomization until disease progression or death, whatever occurs first.

SECONDARY OUTCOMES:
failure of treatment strategy | Until end of follow up (24 months after randomization)
  Time from randomization until failure (death/ progression) of treatment strategy
Progression-free survival of re-induction | From start of re-induction therapy until progress or end of follow-up (24 months after randomization)
  Progression-free survival during re-induction therapy
Objective response after 12 weeks of induction chemotherapy | 12 weeks after start of induction chemotherapy
  Objective response after 12 weeks of induction chemotherapy
Objective best response during maintenance and re-induction | Start of maintenance- until end of re-inductin therapy (expected average of 8 months)
  Objective best response during maintenance and re-induction
Overall survival | Until end of follow-up (24 months after randomization)
  Overall survival measured from time of randomization and from time of registration
Safety | Until end of follow-up (24 months after randomization)
  Overall safety
Health and skin related Quality of life | Until end of follow-up (24 months after randomization)
  Health and skin related Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Trarbach, Dr. med., Principal Investigator — Zentrum für Tumorbiologie und Integrative Medizin, Klinikum Wilhelmshaven
Locations (2):
- Germany (2):
  - St.-Antonius-Hospital Eschweiler, Eschweiler
  - Zentrum für Tumorbiologie und Integrative Medizin, Klinikum Wilhelmshaven, Wilhelmshaven

REFERENCES:
- [Derived] Stahler A, Modest DP, Stintzing S, Borelli B, Keller T, Held S, Fischer von Weikersthal L, Muller L, Graeven U, Decker T, Heintges T, Kahl C, Hoppe B, Kiani A, Kaiser F, Schwaner I, Fruehauf S, Karthaus M, Trarbach T, Klauschen F, Horst D, Cremolini C, Heinemann V. Individual Patient Data Meta-Analysis of Consensus Molecular Subtypes as Biomarkers of First-Line Treatment in RAS Wild-Type Metastatic Colorectal Cancer. J Clin Oncol. 2026 Jan;44(1):31-41. doi: 10.1200/JCO-25-00596. Epub 2025 Nov 18. PMID 41252656
- [Derived] Ballhausen A, Swoboda S, Horst D, Fruehauf S, Graeven U, Muller L, Trarbach T, Fischer von Weikersthal L, Goekkurt E, Heinemann V, Kasper S, Kurreck A, Alig AHS, Reinacher-Schick AC, Bullinger L, Stahler A, Stintzing S, Jarosch A, Modest DP. Spatial Tumor Immune Microenvironment as a Prognostic and Predictive Biomarker in Anti-EGFR-Based Maintenance for RAS wt Metastatic CRC-The PanaMa (AIO KRK0212) Trial. Clin Cancer Res. 2025 Oct 1;31(19):4049-4058. doi: 10.1158/1078-0432.CCR-25-0879. PMID 40736443
- [Derived] Stahler A, Karthaus M, Fruehauf S, Graeven U, Muller L, Fischer von Weikersthal L, Caca K, Goekkurt E, Ballhausen A, Sommerhauser G, Alig AHS, Held S, Jarosch A, Horst D, Reinacher-Schick A, Kasper S, Heinemann V, Stintzing S, Trarbach T, Modest DP. Panitumumab plus 5-fluorouracil and folinic acid or 5-fluorouracil and folinic acid alone as maintenance therapy in RAS wild-type metastatic colorectal cancer (PanaMa, AIO KRK 0212): final efficacy analysis of a randomised, open-label, phase 2 trial. EClinicalMedicine. 2024 Dec 16;79:103004. doi: 10.1016/j.eclinm.2024.103004. eCollection 2025 Jan. PMID 39802302
- [Derived] Stahler A, Kind AJ, Sers C, Mamlouk S, Muller L, Karthaus M, Fruehauf S, Graeven U, Fischer von Weikersthal L, Sommerhauser G, Kasper S, Hoppe B, Kurreck A, Held S, Heinemann V, Horst D, Jarosch A, Stintzing S, Trarbach T, Modest DP. Negative Hyperselection of Resistance Mutations for Panitumumab Maintenance in RAS Wild-Type Metastatic Colorectal Cancer (PanaMa Phase II Trial, AIO KRK 0212). Clin Cancer Res. 2024 Apr 1;30(7):1256-1263. doi: 10.1158/1078-0432.CCR-23-3023. PMID 38289994
- [Derived] Ballhausen A, Karthaus M, Fruehauf S, Graeven U, Muller L, Konig AO, von Weikersthal LF, Sommerhauser G, Alig AHS, Goekkurt E, Meyer-Knees JW, Kurreck A, Stahler A, Held S, Kasper S, Heinrich K, Heinemann V, Stintzing S, Trarbach T, Modest DP. Health-related quality of life in patients with RAS wild-type metastatic colorectal cancer treated with fluorouracil and folinic acid with or without panitumumab as maintenance therapy: a prespecified secondary analysis of the PanaMa (AIO KRK 0212) trial. Eur J Cancer. 2023 Sep;190:112955. doi: 10.1016/j.ejca.2023.112955. Epub 2023 Jun 28. PMID 37454537
- [Derived] Stahler A, Hoppe B, Na IK, Keilholz L, Muller L, Karthaus M, Fruehauf S, Graeven U, Fischer von Weikersthal L, Goekkurt E, Kasper S, Kind AJ, Kurreck A, Alig AHS, Held S, Reinacher-Schick A, Heinemann V, Horst D, Jarosch A, Stintzing S, Trarbach T, Modest DP. Consensus Molecular Subtypes as Biomarkers of Fluorouracil and Folinic Acid Maintenance Therapy With or Without Panitumumab in RAS Wild-Type Metastatic Colorectal Cancer (PanaMa, AIO KRK 0212). J Clin Oncol. 2023 Jun 1;41(16):2975-2987. doi: 10.1200/JCO.22.02582. Epub 2023 Apr 5. PMID 37018649
- [Derived] Sommerhauser G, Kurreck A, Beck A, Fehrenbach U, Karthaus M, Fruehauf S, Graeven U, Mueller L, Koenig AO, V Weikersthal LF, Goekkurt E, Haas S, Stahler A, Heinemann V, Held S, Alig AHS, Kasper S, Stintzing S, Trarbach T, Modest DP. Depth of response of induction therapy and consecutive maintenance treatment in patients with RAS wild-type metastatic colorectal cancer: An analysis of the PanaMa trial (AIO KRK 0212). Eur J Cancer. 2023 Jan;178:37-48. doi: 10.1016/j.ejca.2022.09.011. Epub 2022 Oct 25. PMID 36399909
- [Derived] Modest DP, Karthaus M, Fruehauf S, Graeven U, Muller L, Konig AO, Fischer von Weikersthal L, Caca K, Kretzschmar A, Goekkurt E, Haas S, Kurreck A, Stahler A, Held S, Jarosch A, Horst D, Reinacher-Schick A, Kasper S, Heinemann V, Stintzing S, Trarbach T. Panitumumab Plus Fluorouracil and Folinic Acid Versus Fluorouracil and Folinic Acid Alone as Maintenance Therapy in RAS Wild-Type Metastatic Colorectal Cancer: The Randomized PANAMA Trial (AIO KRK 0212). J Clin Oncol. 2022 Jan 1;40(1):72-82. doi: 10.1200/JCO.21.01332. Epub 2021 Sep 17. PMID 34533973
- See also: Homepage of the AIO (Arbeitsgemeinschaft Internistische Onkologie in der Deutschen Krebsgesellschaft e.V.) — http://www.aio-portal.de